CLINICAL TRIAL: NCT02894736
Title: Home-administered Transcranial Direct Current Stimulation (tDCS) Treatment for Depression
Brief Title: Home-Administered Trial of Direct Current Stimulation
Acronym: HAT-DCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC15010
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active tDCS (Experimental): Soterix tDCS machine is used to administer active stimulation
  Interventions: Device: Soterix tDCS machine

INTERVENTIONS:
Device: Soterix tDCS machine — Soterix tDCS machine - miniCT supervised neuromodulation system

SUMMARY:
Transcranial Direct Current Stimulation (tDCS) is a novel non-invasive brain stimulation treatment that is effective with no significant side effects. It can potentially be self-administered by patients in their own homes with remote monitoring, substantially reducing treatment costs and increasing accessibility, including to remote areas. This study will evaluate the feasibility and efficacy of home-administered tDCS treatment for depression.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets criteria for a DSM-IV Major Depressive Episode, lasting more than 4 weeks
* Total MADRS score ≥ 20

Exclusion Criteria:

* Diagnosis of any DSM-IV psychotic disorder
* History of drug or alcohol abuse or dependence in the preceding 3 months
* High suicide risk
* Clinically defined neurological disorder or insult
* Metal in the cranium or skull defects
* Skin lesions on the scalp (e.g. cuts, abrasions, rashes) at the proposed electrode sites
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Alonzo, BSc(Hons)/BA, PhD, Principal Investigator — University of New South Wales / Black Dog Institute
Locations (1):
- Black Dog Institute, Randwick, Sydney, New South Wales, Australia